CLINICAL TRIAL: NCT04607564
Title: Formative Research and Development of a Sexual Violence Prevention Intervention for South African Higher Education Institutions
Brief Title: Pilot Study of the Ntombi Vimbela Sexual Violence Intervention Among Female Tertiary Students in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Mercilene Machisa, Specialist Scientist, Medical Research Council, South Africa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC002/2/2018
Record Dates: First submitted 2020-10-01; First posted 2020-10-29 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Sexual Violence

STUDY DESIGN:
Intervention Model Description: This is a pilot and feasibility study where sites are conveniently selected and the recruitment of participants is by invitation and non-randomised. All participants will receive the Ntombi Vimbela intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No comparison pilot group (Experimental): Attendance at ten Ntombi Vimbela workshops running for a total 35 hours over six weeks.
  Interventions: Other: Ntombi Vimbela! intervention

INTERVENTIONS:
Other: Ntombi Vimbela! intervention — Ntombi Vimbela! constitutes a series of ten workshops running for a total 35 hours. The intervention is designed to raise awareness about sexual rights, violence against women and girls and its drivers; sensitise about gender inequality and build more gender equitable beliefs; sensitise about sexual assault; equip participants with skills to assess and act in situations where there is a high risk of sexual assault; build resilience and skills to withstand social and material pressures in college or university ; enable utilisation of health, psycho-social services and access to justice for survivors; enhance communication skills and building healthy sexual relationships; promote mental health and coping and build empathy towards survivors.

SUMMARY:
The pilot study aims to test the acceptability of content, feasibility of delivery methods and preliminary assessment of outcomes from the implementation of the Ntombi Vimbela intervention with volunteer groups of female first year students at eight South African higher education campuses. Data to inform the different objectives will be collected from participants at different time points. A baseline questionnaire was administered at the beginning of the Ntombi Vimbela workshops. Qualitative data to provide evidence about the workshop content and relevance was collected using participant end of workshop evaluation forms and end of intervention delivery focus group discussions.Feasibility data was collected through research team observations, facilitator debriefings and end of intervention delivery workshop One year post-implementation data which provides evidence of preliminary impact has commenced which includes a survey and in-depth interviews with participants.

DETAILED DESCRIPTION:
Facilitator recruitment and training: The intervention piloting will be conducted in eight selected campuses. In each campus, three facilitators will be recruited through a process involving advertisements, applications, screening and interview. This makes a total of nine facilitators. The criteria for facilitators will be full time female students, between the ages of 25 and 30 years of age, enrolled at the institution for at least one year. Facilitators will be trained by the lead researchers to recruit participants and run intervention with groups of participants. The facilitator training will be conducted by the lead researchers over a duration of seven days. The training will cover the intervention content, participatory delivery protocol, group facilitation techniques, dynamics of co-facilitation and problem-solving techniques.

Project marketing and participant recruitment: First posters about the study will be put up in lecture rooms, residences and central meeting points at selected campuses. Posters will have information which will include the study aims, participation criteria and contact details of the project managers. Facilitators will also approach students, share the study information and invite them to participate. The Student Support managers will also assist in publicising the project as they conduct their normal duties. In each institution, 20 students will be recruited to participate in the intervention. To be eligible to participate, a student has to be female, aged 18-30 years and a full-time student at the college. At the final stage of recruitment, participants will receive the written project information leaflet and will be required to give written consent prior to participation. Participants will also be required to provide their contact details which will be used to communicate project activities.

Participant assessments and feedback: Prior to participating in the programme, participants will be required to complete a short baseline questionnaire that includes measures of their background data, gender attitudes, perceptions of sexual violence, violence exposures, knowledge or use of campus support services or other forms of support (informal and formal). The same tool used at baseline will be used at 1 year post-implementation of workshops to assess any changes in knowledge, attitudes and behaviour. In compliance to the COVID-19 regulations the researchers will contact participants and invite them to participate remotely. A survey link will be sent to them which they will use to complete the questionnaire. For the qualitative follow up component, researchers will systemically sample half of the participants at each site and invite them to participate in telephonic in-depth interviews. On agreed days and times, researchers will conduct the telephonic interview using a structured guide. All interviews will be audio-recorded, transcribed verbatim and translated into English in preparation for analysis. The assessments are solely for the purpose of assessing the acceptability and feasibility of the intervention and impact evaluation.

Facilitator support, debriefing and feedback: During the implementation of the programme, facilitators will be expected to fill attendance records, collect filled participant evaluation forms and compile session reports. Attendance record will allow us to ascertain whether workshop attendance gets sustained throughout the four sessions. Facilitators will use session reports to document challenges encountered and how those were resolved; which exercises worked well and which did not; what do they think could be done to make the exercises work better. Each facilitator will be expected to attend a weekly two-hour face to face debriefing and planning meeting chaired by the lead researchers. The debriefing sessions will be used to engage with the participant evaluations and as a means of getting facilitator feedback relating to intervention delivery. Facilitators will also be expected to request the inputs of the project manager when dealing with any challenges in implementation. In closing the implementation, in-depth one-on-one interviews will be conducted with facilitators on their experiences of delivering the intervention, reflecting on similar issues as are observed for participants. A focus group discussion will also be conducted with all facilitators to allow them to discuss in detail amongst themselves the challenges, successes and suggest improvements to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female students,
* Ages 18-30 years
* First year students

Exclusion Criteria:

* Female students Ages 31+
* Post graduate students
* Students enrolled for at institution for more than 1 year

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in personal gender beliefs from baseline | 1 year
  Assessed by a summative score from 8 items of the Gender Equitable Men Scale Score . Scale items include "I think that a woman should obey her husband. I think that a man should have the final say in all family matters I think that men should share the work around the house with women such as doing dishes, cleaning and cooking. I think that if someone insults a man he should be prepared to physically fight to defend his honour.I think that if a wife does something wrong her husband has the right to punish her. I think that there are times when a woman deserves to be beaten.I think that it is possible for a woman to be raped by her husband. I think that people should be treated the same whether they are male or female" Possible responses are in likert scale : 1=strongly agree, 2=agree, 3=disagree, 4=strongly disagree
Change in sexual self efficacy from baseline | 1 year
  Assessed by a summative score from 12 items of the Sexual Efficacy Scale. Scale items include "Would you be able to use a condom every time you have sex?Would you be able to buy your own condoms or contraception? Would you be able to refuse to have sex without condom? Would you be able to talk to your partner about his previous sexual activities? Would you be able to talk about using contraception with your partner? Would you be able to talk about using condoms with your partner? Would you be able to tell your partner how he should treat you sexually and the kind of sex you like? Would be able to refuse sex with your partner? Would be able to refuse sex with someone whom you want to date again ? Would be able to refuse sex with someone whom you want to fall in love with you? Would you be able to refuse to do something sexual if you didn't want it? Would you be able to meet your own sexual needs through masturbation" Possible responses are 1=No ; 2=Probably not; 3= Probably; 4=Yes
Past year incidence of non-partner rape | 1 year
  Assessed using a modified version of the World Health Organisation's Domestic Violence Questionnaire. Items include "How many times were you forced by someone who was not your boyfriend/husband to have oral sex? How many times were you forced by someone who was not your boyfriend/husband to have penetrative sex? How many times were you forced to have sex with a man when you didn't want to but you were too drunk or drugged to stop it? How many times were you forced to have sex with more than one man at the same time?" Possible responses 1=Never, 2=Once, 3=More than one time Has this happened in the past 12 months? Possible response Yes/No
Past year incidence of partner sexual violence | 1 year
  Assessed using a modified version of the World Health Organisation's Domestic Violence Questionnaire . Items include "Has a current or previous husband or boyfriend ever forced you to do something sexual that you found degrading or humiliating? Did this happen many times, a few times, once or did it not happen? Have you ever had sex with a boyfriend/husband when you didn't want to because he physically forced or threatened or pressured you? Possible responses 1=Never, 2=Once, 3=More than one time Has this happened in the past 12 months? Possible responses Yes/No
Self defence self efficacy | 1 year
  Assessed by a summative score of 8 adapted items of Self defence Self efficacy scales. Example of items include "If I sense anything about a man that makes me uncomfortable, I'm able to avoid being alone with him.If my date refused to stop after I told him to, I wouldn't know what I could do to make him stop. I know a number of basic hand strike self defense moves e.g straight punch, knife hand, hammer fist that I would be able to use if anyone tried to rape me. I know a number of basic kicking self defense moves e.g front or back kicks that I would be able to use if anyone tried to rape me. I know a number of basic elbow self defense moves that I would be able to use if anyone tried to rape me. I know a number of basic wrist release self defense moves that I would be able to use if anyone tried to rape me. Possible responses 1=strongly agree, 2=agree, 3=disagree, 4=strongly disagree

SECONDARY OUTCOMES:
Change in mental health from baseline | 1 year
  Change in depression scores summed from responses to 20 items from the Centre for Epidemiologic Studies Depression (CES-D) Scale. 21+ cut off score used to indicate depressive symptoms
Change in self esteem from baseline | 1 year
  Assessed by a summative score of 10 items of the Rosenberg's Self esteem scale. Scale items include "I feel good about myself. I feel satisfied with the way my body looks right now. I am pleased with my appearance right now.
  I am satisfied with my weight right now. I feel sexually unattractive. I am worried about what other students and people think of me. I am able to do things as well as most other people. I feel that others respect and admire me.
  I can do just about anything I set my mind to do. I have great faith in the future" Possible responses in Likert Scale i.e strongly agree, agree, disagree, strongly disagree
Change in rape myth acceptance from baseline | 1 year
  Assessed by a summative score of 14 adapted items of the Illinois Rape Myths Scale. Example of scale items include " I think that when a woman is raped, she is usually to blame for putting herself in that situation.I think that women are raped because they lead men on. I think that if a woman behaves like a slut, she will be raped. I think that if a woman dresses in short and skimpy clothes, she is inviting men to rape her. I think that if a woman goes to a room alone with a man at a party, she is to blame if she gets raped. I think that women get raped because they do not say NO clearly. I think that if a woman doesn't verbally resist it's not rape. I think that if a woman doesn't physically resist or fight back, it's not rape.I think when men rape, it is because they are unable to control their strong desire for sex. I think that it cant be rape if both the man and woman are drunk. Possible responses are in Likert scale i.e 1=Strongly agree, 2=agree, 3=disagree, 4=strongly disagree
Change in emotional help seeking behaviours from baseline | 1 year
  Assessed by a summative score of a scale of six items i.e When feeling sad, disappointed or frustrated have you sought help from older relatives? When feeling sad, disappointed or frustrated have you sought professional counselling e.g from a social worker or psychologist? When feeling sad, disappointed or frustrated have you sought help through family meetings? When feeling sad, disappointed or frustrated have you sought help from the student support servcies ? When feeling sad, disappointed or frustrated have you sought help from a doctor? When feeling sad, disappointed or frustrated have you turned to prayer or sought help from religious person? When feeling sad, disappointed or frustrated have you sought help from a local non governmental organisation " Possible responses 0=No; 1=Yes

CONTACTS AND LOCATIONS:
Overall Officials: Mercilene Machisa, PhD, Principal Investigator — Medical Research Council, South Africa; Rachel Jewkes, MBBS, Study Director — Medical Research Council, South Africa
Locations (6):
- South Africa (6):
  - University of Fort Hare, Alice, Eastern Cape
  - South West Gauteng TVET College, Johannesburg, Gauteng
  - Elangeni TVET College, Pinetown, KwaZulu-Natal
  - University of Limpopo, Mankweng, Limpopo
  - Ehlanzeni TVET College, Mbombela
  - Lovedale TVET College, Qonce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Machisa MT, Mahlangu P, Chirwa E, Nunze N, Sikweyiya Y, Dartnall E, Pillay M, Jewkes R. Ntombi Vimbela! Sexual violence risk reduction intervention: pre and one-year post assessments from a single arm pilot feasibility study among female students in South Africa. BMC Public Health. 2023 Jun 27;23(1):1242. doi: 10.1186/s12889-023-16149-x. PMID 37370055